CLINICAL TRIAL: NCT06142474
Title: The Potential Beneficial Effects of SGLT2 Inhibitors in Patients With Acute Decompensated Heart Failure During Ventilator Weaning: a Prospective Multicenter Cohort Study.
Brief Title: SGLT2 Inhibitors in Patients With ADHF During Ventilator Weaning
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Chih Fan Yeh, MD, PhD, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209061MINA
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure Acute; Ventilator Lung
Keywords: Heart Failure Acute; Ventilator
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; empagliflozin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acute decompensated HF Patients (No Intervention): acute decompensated HF Patients 2：1，have 50 Patients control and 100 Patients randomly assigned empagliflozin or dapagliflozin
- empagliflozin 10mg (Experimental): acute decompensated HF Patients 2：1,have 50 Patients control and 100 Patients randomly assigned empagliflozin or dapagliflozin ,3 days before ventilator weaning in a ratio of 1:1.empagliflozin 10 mg once daily
  Interventions: Drug: SGLT2 inhibitor
- dapagliflozin 10mg (Experimental): acute decompensated HF Patients 2：1,have 50 Patients control and 100 Patients randomly assigned empagliflozin or dapagliflozin ,3 days before ventilator weaning in a ratio of 2:1. dapagliflozin 10 mg once daily
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Patients with acute decompensated HF will be open-label randomly assigned to be treated with or without SGLT2 inhibitors (either empagliflozin 10 mg once daily or dapagliflozin 10 mg once daily) 3 days before ventilator weaning in a ratio of 2:1. If the patients are allocated to SGLT2i treatment group, they will be further randomized equally to either empagliflozin- or dapagliflozin-treated group
  Other Names: Empagliflozin and dapagliflozin
  Arms: dapagliflozin 10mg; empagliflozin 10mg

SUMMARY:
This study will explore the potential benefits of sodium-glucose cotransporter 2 (SGLT2) inhibitors in preventing cardiac ischemia and cardiopulmonary edema in patients with acute decompensated heart failure during weaning from ventilators.

DETAILED DESCRIPTION:
Patients with acute decompensated HF will be open-label randomly assigned to be treated with or without SGLT2 inhibitors (either empagliflozin 10 mg once daily or dapagliflozin 10 mg once daily) 3 days before ventilator weaning in a ratio of 2:1. If the patients are allocated to SGLT2i treatment group, they will be further randomized equally to either empagliflozin- or dapagliflozin-treated group. A series of examination will be performed to detect weaning-induced cardiac ischemia and weaning-induced cardiopulmonary edema, including electrocardiography, chest X-ray, echocardiography, and biomarkers.

Echocardiography Transthoracic echocardiography (TTE) will be performed by a trained operator at several time points: (1) before SBT and SGLT2i initiation; (2) during SBT trial just after initiating SGLT2 inhibitor; (3) during SBT trial 3 days after initiation of SGLT2 inhibitor; (4) within 24 hrs after extubation; (5) 7-10 days after extubation; (6) 90±7 days after extubation.

Biomarkers NT-proBNP, plasma protein, high-sensitive cardiac troponin T, and hemoglobin level will be checked at several time points: (1) before spontaneous breathing trial (SBT), (2) during SBT trial (at least 10 mins after the initiation of SBT) just after initiating SGLT2 inhibitor; (3) during SBT (at least 10 mins after the initiation of SBT) trial 3 days after SGLT2 inhibitor; (4) within 24 hrs after extubation; (5) 7~10 days after extubation; (5) 90±7 days after extubation. We will also check arterial blood gas analyses at the end of SBT trial just after initiating SGLT2 inhibitor and 3 days after SGLT2 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥20 years
2. Currently hospitalized for the primary diagnosis of acute HF (de novo or decompensated chronic HF) in HFrEF patients (LVEF≤40%)
3. Meet the stabilization criteria:

   A. Systolic BP ≥100mm Hg and no symptoms of hypotension in the preceding 6 hours B. No increase in i.v. diuretic dose for 6 hours prior to randomization C. No i.v. vasodilators including nitrates within the last 6 hours prior to randomization D. No i.v. inotropic drugs for 24 hours prior to randomization
4. Elevated N-terminal proB-type natriuretic peptide (NT-proBNP) or BNP:

   A. Without atrial fibrillation (AF): NT-proBNP ≥1600 pg/mL or BNP ≥400 pg/mL B. With AF: NT-proBNP ≥2400 pg/mL or BNP ≥600 pg/mL
5. Patients were intubated for at least 24 hour with ventilator settings allowing to initiate the weaning process [SpO2 > 90% or PaO2/FiO2 ≥ 150 mmHg with a fraction of inspired oxygen (FiO2) ≤ 40% and a positive end-expiratory pressure (PEEP) ≤ 8 cmH2O].

Exclusion Criteria:

1. Decision to withdraw life support
2. Cardiogenic shock
3. Hospitalization for HF (HHF) triggered by acute myocardial infarction (AMI) or pulmonary embolism
4. Planned or previous (within 30 days) cardiovascular revascularization or major cardiac surgery/intervention/device implantation
5. Prior acute coronary syndrome, AMI, stroke or transient ischemic accident within 90 days
6. Estimated glomerular filtration rate (eGFR) of less than 30 ml per minute per 1.73 m2 of body-surface area
7. Type 1 diabetes mellitus
8. Poorly controlled type 2 diabetes mellitus (a glycated hemoglobin level above 10.5%)
9. Uncontrolled urinary tract infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2030-10-09 (Estimated); Study Completion 2030-10-09 (Estimated)

PRIMARY OUTCOMES:
Composite of weaning failure, recurrent pulmonary edema, and cardiovascular/non-cardiovascular mortality. | 90 days
  Weaning failure is defined that patient is reintubated within 7 days following extubation, irrespective of the use of noninvasive ventilation

SECONDARY OUTCOMES:
Components of the primary endpoint | 90 days
  Weaning failure, recurrent pulmonary edema, and cardiovascular/non-cardiovascular mortality.
Diuretic response | after 15 and 30 days of treatment
  Any poor response to diuretics
Change in NT-proBNP level | over 30 days of treatment
  Difference between 30 days and baseline
Occurrence of chronic dialysis or renal transplant or significant, sustained reduction of estimated glomerular filtration rate | 90 days
  Dialysis, renal transplant and eGFR
The therapeutic effect by different SGLT2i on components of the primary endpoint. | 90 days
  Empagliflozin vs Dapagliflozin

OTHER OUTCOMES:
Safety parameters | 30 days
  Markers of volume depletion, hypotension and acute renal failure

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- [Background] Spertus JA, Birmingham MC, Nassif M, Damaraju CV, Abbate A, Butler J, Lanfear DE, Lingvay I, Kosiborod MN, Januzzi JL. The SGLT2 inhibitor canagliflozin in heart failure: the CHIEF-HF remote, patient-centered randomized trial. Nat Med. 2022 Apr;28(4):809-813. doi: 10.1038/s41591-022-01703-8. Epub 2022 Feb 28. PMID 35228753
- [Background] Solomon SD, McMurray JJV, Claggett B, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Jhund PS, Belohlavek J, Chiang CE, Borleffs CJW, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer-Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Saraiva JFK, Tereshchenko SN, Thierer J, Vaduganathan M, Vardeny O, Verma S, Pham VN, Wilderang U, Zaozerska N, Bachus E, Lindholm D, Petersson M, Langkilde AM; DELIVER Trial Committees and Investigators. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1089-1098. doi: 10.1056/NEJMoa2206286. Epub 2022 Aug 27. PMID 36027570
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503